CLINICAL TRIAL: NCT00612560
Title: Flaxseed vs. Aromatase Inhibitors: Breast Tumor Characteristics and Prognosis
Brief Title: Flaxseed, Aromatase Inhibitors and Breast Tumor Characteristics
Acronym: FABrC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: I 99507; I99507; R21AT004024-01 (NIH); NCT00635908 (obsolete NCT alias)
Record Dates: First submitted 2008-02-07; First posted 2008-02-11 (Estimated); Results first posted 2017-08-16 (Actual); Last update posted 2017-10-12 (Actual); Status verified 2017-09

CONDITIONS: Breast Cancer
Keywords: breast neoplasms; phytoestrogens; tumor characteristics; proliferation; apoptosis; estrogen receptor; HER2
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole; Linseed Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 2 (Experimental): Flaxseed 25 mg per day and 1 placebo pill per day
  Interventions: Dietary Supplement: flaxseed
- 3 (Experimental): 25 mg flaxseed per day and 1 mg anastrozole pill per day
  Interventions: Drug: Anastrozole; Dietary Supplement: flaxseed
- 4 (Placebo Comparator): Placebo pill 1 per day
  Interventions: Drug: Placebo
- 1 (Experimental): Anastrozole 1 mg pill per day
  Interventions: Drug: Anastrozole

INTERVENTIONS:
Drug: Anastrozole — 1 mg per day
  Other Names: Arimidex
  Arms: 1; 3
Dietary Supplement: flaxseed — 25 g per day ground
  Arms: 2; 3
Drug: Placebo — Placebo pill 1 per day
  Arms: 4

SUMMARY:
The proposed study plans to examine the effect of flaxseed consumption, a phytoestrogen rich food, compared to aromatase inhibitors as a complementary approach to treating estrogen receptor positive breast cancer, as well as the effect of combined flaxseed and aromatase inhibitor therapy on breast cancer treatment. Because of the increasing use of both complementary and alternative approaches to treatment, and the use of aromatase inhibitors in the treatment of breast cancer, the proposed study has potential to provide important clinical information about the effect of foods high in phytoestrogens on a common endocrine therapy used in breast cancer.

DETAILED DESCRIPTION:
Although the 10 year survival rate for women with early stage breast cancer is very good, distant recurrence is still a serious concern, especially for estrogen receptor positive women. Consequently, breast cancer survivors are interested in therapies that might improve their recurrence free survival (RFS). Used in postmenopausal women, aromatase inhibitors (AI) block the peripheral conversion of androgens to estrogen, effectively lowering the estradiol available to promote breast tumor proliferation. However, use of AIs is associated with hot flashes, joint pain, bone loss, and an increase in cardiac events. Furthermore, many breast tumors eventually develop resistance to hormonal treatments. Complementary and alternative medicines (CAMs) are widely used by cancer survivors in an attempt to reduce disease recurrence with fewer side effects and potential health benefits, and use is particularly prevalent among breast cancer survivors. Flaxseed (FS) is a commonly available food often consumed as a dietary supplement and is the richest food source of lignans, a phytoestrogen. In experimental models, flaxseed consumption has been shown to exhibit a number of activities that suggest a potential benefit of flaxseed in the adjuvant setting. However, the majority of human studies investigating the biologic effects of flaxseed have involved healthy women. There is a paucity of clinical data regarding the efficacy and safety of use of flaxseed among women with breast cancer, especially among those receiving AIs. Because the phytoestrogens in flaxseed can influence many of the same biologic pathways affected by hormonal agents, diet-drug interactions are possible. Additionally, it is possible flaxseed could act through growth and signaling pathways, modifying the development of endocrine resistance. Potential synergistic or antagonistic effects between flaxseed and antiestrogens are of particular interest given the increasing use of AIs to treat postmenopausal women with hormone responsive disease. We propose to conduct a pilot 2x2 factorial randomized intervention study between tumor biopsy and resection, in postmenopausal women diagnosed with ER positive breast cancer, to assess the effects of flaxseed and AI on a number of steroid hormone and tumor-related characteristics associated with long-term survival, and to investigate the potential interaction between flaxseed and AI on tumor expression of Ki-67, caspase, ERα, ERβ, PgR, HER2, IGF1, IGFIR. The pre-surgical setting offers a unique opportunity to rapidly obtain information on intervention related effects on growth factor and signaling pathways related to tumor characteristics in a short time period without the interference of other treatments. We hypothesize that both flaxseed and AI interventions will independently favorably affect growth factor and signaling pathway protein expression resulting in reduced tumor proliferation and increased apoptosis. We further hypothesize that these improvements will be reflected in improved recurrence scores as estimated by the Mammostrat antibody panel (Applied Genomics Incorporated). The proposed study will provide important clinical data for future dietary intervention studies involving phytoestrogen lignans from flaxseed.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 85 years
* Postmenopausal status defined as: no menstrual cycle in the past 12 months hysterectomy with bilateral oophorectomy hysterectomy with intact ovaries if age > 55 years
* Newly diagnosed with incident, primary, invasive, estrogen receptor positive clinical stage II or lower breast cancer
* ECOG performance status of 1 or less
* Willingness to comply with study guidelines and procedures
* Willingness and ability to provide informed consent
* Usual consumption of soy no more than 1 time per week and willingness to avoid whole soy foods or concentrated soy sources (soy milk, tofu, substitute meat products, meal replacement bars) during the intervention period
* Willingness to avoid herbal and dietary supplements (not including vitamins), aspirin, and ibuprofen during the intervention period
* No competing neoadjuvant or chemotherapy treatment
* Time between pre-surgical visit and surgery must be at least 2 weeks
* No chemotherapy in the past 12 months

Exclusion Criteria:

* Inability to read and write English
* Previous invasive breast cancer
* Insulin dependent Type I or II diabetes diagnosed by physician
* History of coagulopathy, thrombocytopenia, or bleeding disorder
* Current (past 30 days) regular (at least once per week) use of reproductive hormone therapy, Tamoxifen, aromatase inhibitors, or other estrogen inhibitors, flaxseed, or antibiotics
* Current chemotherapy or neoadjuvant chemotherapy
* Allergies to flaxseed, nuts, or other seeds
* Renal dysfunction defined as creatinine > 1.5 mg/dl
* History of Crohns' disease, ulcerative colitis, irritable bowel syndrome, celiac sprue, or other malabsorption syndrome, diverticulitis, diverticulosis, or other bowel diagnosis which, in the opinion of the breast surgeon, would contraindicate large doses of dietary fiber or would impair nutrient absorption
* Current, regular (more than once weekly) use of prescription blood-thinning agents including coumadin, heparin and heparin related drugs, clopidogrel bisulfate

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2007-11; Primary Completion 2011-01 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tracey L O'Connor, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

REFERENCES:
- [Derived] McCann SE, Edge SB, Hicks DG, Thompson LU, Morrison CD, Fetterly G, Andrews C, Clark K, Wilton J, Kulkarni S. A pilot study comparing the effect of flaxseed, aromatase inhibitor, and the combination on breast tumor biomarkers. Nutr Cancer. 2014;66(4):566-75. doi: 10.1080/01635581.2014.894097. Epub 2014 Mar 26. PMID 24669750

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A - Flaxseed & Active Anastrazole: 25 mg flaxseed per day and 1 mg anastrozole pill per day
  Anastrozole: 1 mg per day
  flaxseed: 25 g per day ground
- Arm B - Flaxseed: Flaxseed 25 mg per day and 1 placebo pill per day
  flaxseed: 25 g per day ground
- Arm C - Anastrozole: Anastrozole 1 mg pill per day
  Anastrozole: 1 mg per day
- Arm D - Placebo: Placebo pill 1 per day
  Placebo: Placebo pill 1 per day
Period: Overall Study
Arm/Group | Arm A - Flaxseed & Active Anastrazole | Arm B - Flaxseed | Arm C - Anastrozole | Arm D - Placebo
Started | 7 | 7 | 8 | 6
Completed | 7 | 7 | 8 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All treated and eligible patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A - Flaxseed & Active Anastrazole | Arm B - Flaxseed | Arm C - Anastrozole | Arm D - Placebo | Total
Number analyzed (Participants) | 7 | 7 | 8 | 6 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 6 | 4 | 3 | 16
  >=65 years | 4 | 1 | 4 | 3 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (8.5) | 58 (7.5) | 65 (6.6) | 64 (7.6) | 62 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 8 | 6 | 28
  Male | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 1
  White | 7 | 6 | 8 | 6 | 27
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Expression of Estrogen Receptor (ER-beta)
Description: Mean percentage of cells expressing estrogen receptor (ER-beta)
Time Frame: Biopsy/Week 1 and Surgical Resection/Week 2
Population: All treated and eligible patients with a large enough of a sample for analysis
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Arm A - Flaxseed & Active Anastrazole | Arm B - Flaxseed | Arm C - Anastrozole | Arm D - Placebo
Number analyzed (Participants) | 7 | 6 | 4 | 6
percentage of cells
  Biopsy: number analyzed (Participants) | 7 | 6 | 4 | 5
  Biopsy | 67.1 (17.0) | 63.3 (10.3) | 45.0 (23.8) | 62.0 (13.0)
  Surgical resection: number analyzed (Participants) | 7 | 6 | 3 | 6
  Surgical resection | 45.7 (28.8) | 56.7 (23.4) | 46.7 (32.1) | 70 (30.9)

2. Primary Outcome: Progesterone Receptor (PR) Expression
Description: Mean percentage of cells expressing PR
Time Frame: Biopsy/Week 1 and Surgical Resection/Week 2
Population: All treated and eligible patients with a large enough of a sample for analysis
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Arm A - Flaxseed & Active Anastrazole | Arm B - Flaxseed | Arm C - Anastrozole | Arm D - Placebo
Number analyzed (Participants) | 2 | 5 | 2 | 4
percentage of cells
  Biopsy: number analyzed (Participants) | 2 | 5 | 1 | 4
  Biopsy | 4 (1.4) | 3.5 (0.7) | 2 | 4.7 (0.5)
  Surgical resection: number analyzed (Participants) | 2 | 5 | 2 | 2
  Surgical resection | 4.5 (0.7) | 2.4 (1.1) | 1 (1.4) | 3.5 (2.1)

3. Primary Outcome: Human Epidermal Growth Factor Receptor 2 (Her2) Expression
Description: Mean percentage of cells expressing human epidermal growth factor receptor 2 (Her2)
Time Frame: Biopsy/Week 1 and Surgical Resection/Week 2
Population: All treated and eligible patients with a large enough of a sample for analysis.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Arm A - Flaxseed & Active Anastrazole | Arm B - Flaxseed | Arm C - Anastrozole | Arm D - Placebo
Number analyzed (Participants) | 2 | 4 | 2 | 2
percentage of cells
  Biopsy: number analyzed (Participants) | 2 | 1 | 0 | 2
  Biopsy | 15 (7.0) | 40 |  | 55 (63.6)
  Surgical resection: number analyzed (Participants) | 2 | 4 | 2 | 1
  Surgical resection | 0 (0) | 17.5 (16.6) | 17.5 (17.7) | 30

4. Secondary Outcome: Growth Hormone Serum Levels IGF-1
Description: Mean serum level IGF-1(pg/ml)
Time Frame: Biopsy/Week 1 and Surgical Resection/Week 2
Population: All treated and eligible patients with a large enough of a sample for analysis
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Arm A - Flaxseed & Active Anastrazole | Arm B - Flaxseed | Arm C - Anastrozole | Arm D - Placebo
Number analyzed (Participants) | 6 | 7 | 7 | 6
pg/ml
  Biopsy: number analyzed (Participants) | 6 | 7 | 7 | 5
  Biopsy | 887.7 (654.4) | 1044.2 (700.4) | 959.1 (408.6) | 1008.3 (686.7)
  Surgical resection | 938.1 (652.9) | 980.5 (743.2) | 819.8 (334.3) | 880.1 (698.0)

ADVERSE EVENTS:
Arm/Group | Arm A - Flaxseed & Active Anastrazole | Arm B - Flaxseed | Arm C - Anastrozole | Arm D - Placebo
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 1/8 | 0/6
Other Adverse Events (participants affected / at risk) | 6/7 | 6/7 | 5/8 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A - Flaxseed & Active Anastrazole (N=7) | Arm B - Flaxseed (N=7) | Arm C - Anastrozole (N=8) | Arm D - Placebo (N=6)
Breast haematoma (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A - Flaxseed & Active Anastrazole (N=7) | Arm B - Flaxseed (N=7) | Arm C - Anastrozole (N=8) | Arm D - Placebo (N=6)
Palpitations (Cardiac disorders) | 0 (0) | 2 (10) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (6) | 2 (4) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (10) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (8) | 1 (2) | 0 (0) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (2) | 2 (8) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 5 (12) | 4 (14) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (6) | 2 (2) | 1 (2)
Asthenia (General disorders) | 0 (0) | 1 (2) | 3 (3) | 3 (3)
Chills (General disorders) | 0 (0) | 2 (10) | 1 (1) | 1 (1)
Fatigue (General disorders) | 2 (6) | 0 (0) | 3 (7) | 5 (5)
Feeling abnormal (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Feeling cold (General disorders) | 0 (0) | 2 (8) | 1 (1) | 1 (1)
Irritability (General disorders) | 1 (2) | 1 (2) | 2 (2) | 1 (1)
Oedema peripheral (General disorders) | 1 (2) | 1 (2) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (2) | 1 (2) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Mastitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Incision site pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Incision site pruritus (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural vomiting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Weight increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (6) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (2) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (4) | 1 (2) | 2 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 1 (2) | 1 (4) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (2) | 1 (2) | 2 (2) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (6) | 3 (8) | 1 (1) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 1 (2) | 2 (6) | 0 (0) | 3 (3)
Lethargy (Nervous system disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (2) | 2 (4) | 2 (3) | 2 (2)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (2) | 1 (2) | 2 (2) | 1 (1)
Decreased interest (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Depressed mood (Psychiatric disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (1)
Disturbance in sexual arousal (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (2) | 2 (4) | 2 (2) | 2 (2)
Libido decreased (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Loss of libido (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (6) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (4) | 0 (0) | 3 (5)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 3 (8) | 2 (6) | 2 (2) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (4) | 1 (1) | 1 (1)
Hot flush (Vascular disorders) | 2 (4) | 2 (4) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes